CLINICAL TRIAL: NCT02599558
Title: A Pilot Trial of Dietary Therapy Directed by the Esophageal Sponge in the Management of Eosinophilic Esophagitis.
Brief Title: Cytosponge and Dietary Therapy in EoE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey A Alexander, Prinicipal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-004741
Record Dates: First submitted 2015-11-02; First posted 2015-11-06 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Eosinophilic Esophagitis
Keywords: EOE
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cytosponge-directed food reintroduction (Experimental): Subjects will follow the six-food elimination diet per clinical protocol. The cytosponge will be used to monitor the diet at certain timepoints during food reintroduction
  Interventions: Device: Cytosponge

INTERVENTIONS:
Device: Cytosponge — A capsule with a string attached with a sponge inside is swallowed. The string is held without any tension to allow the capsule to move into the stomach. The string will be held for five minutes to allow the capsule to dissolve in the stomach; a round mesh sponge about the size of a quarter is released.
  Other Names: sponge

SUMMARY:
This study is being done to see if the investigators can use only the cytosponge ( A 10 minute, in office procedure that does not require sedation) to replace the 6-10 endoscopies routinely perform during dietary restriction and food reintroduction in EoE?

DETAILED DESCRIPTION:
Dietary Therapy has been shown to be successful in the treatment of adult and pediatric patients with eosinophilic esophagitis Dietary studies were initially reported in children, but the results appear to be similar in adult patients. Elemental diets are successful in 70-95% of patients but are poorly tolerated. A six food elimination diet has been effective in about 70% of adult patients with EoE . In these adult studies skin prick testing was not helpful in predicting which foods would lead to a flare of disease when reintroduced into the diet. Therefore, the current standard of care requires multiple EGDs with esophageal biopsy during the dietary restriction and reintroduction phases of this study. Since the investigators are making lifelong dietary decisions during this process of food reintroduction, it is imperative the investigators be accurate. Unfortunately, these multiple EGDs have significant cost and are invasive procedures with some risk. Moreover, there is significant indirect costs with travel and time off work for the patients and drivers. Previous studies have found the esophageal sponge to be an accurate technique of accessing esophageal eosinophilia in EoE . The sponge is swallowed as a 12 mm capsule on a string. The capsule rapidly dissolves upon entering the stomach and the sponge then expands and can be pulled out the mouth five minutes after ingestion. In previous studies, the procedure was very well tolerated and all patients preferred the sponge to endoscopy.

Therefore the sponge is a well tolerated, inexpensive, very low risk procedure that would be an ideal option to replace EGD esophageal sampling in the evaluation of dietary treatment of EoE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Eosinophilic Esophagitis > than 15 Eos phf and failed to respond to the PPI therapy
* Going through the six food elimination diet or have just completed elimination the six foods: fish, nuts, eggs, soy, wheat, and milk

Exclusion Criteria:

* Clinical evidence of infectious process potentially contributing to dysphagia ( candidiasis, CMV, herpes)
* Other cause of dysphagia identified at endoscopy (e.g. reflux esophagitis, stricture, web, ring, achalasia, esophageal neoplasm)
* Esophageal minimal diameter < 13 mm on structured barium esophagram

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11; Primary Completion 2022-01-08 (Actual); Study Completion 2022-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Alexander, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Alexander JA, Ravi K, Symrk TC, Wu TT, Lavey CJ, Geno D, Johnson AJ, Lennon RJ, Collins MH, Dellon ES, Katzka DA. Use of the Esophageal Sponge in Directing Food Reintroduction in Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2023 Feb;21(2):299-306.e3. doi: 10.1016/j.cgh.2022.05.029. Epub 2022 Jun 10. PMID 35697266
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials
- See also: Pub Med — https://pubmed.ncbi.nlm.nih.gov/35697266/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cytosponge-directed Food Reintroduction
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cytosponge-directed Food Reintroduction
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Histological Remission by Sponge Cytology
Description: Number of subject's sponge cytology to accurately detect histological remission when compared with standard of care EGD (defined as a peak eosinophil count of <15 eos/hpf on endoscopic biopsy)
Time Frame: approximately 4 weeks post food reintroduction
Measure: Count of Participants; unit: Participants
Arm/Group | Cytosponge-directed Food Reintroduction
Number analyzed (Participants) | 22
Participants | 13

2. Secondary Outcome: Eosinophilic Esophagitis Activity Index Patient Reported Outcomes (EEsAI PRO) Score
Description: The EEsAI PRO questionnaire includes items related to the intensity and frequency of dysphagia, the influence of specific food groups on dysphagia symptoms, and other symptoms independent of eating or drinking (ie, heartburn, acid regurgitation, and chest pain). The total EEsAI PRO score ranges from 0 to 100 (higher score indicates worsening symptoms). A PRO < 20 defines asymptomatic EoE
Time Frame: approximately 4 weeks post food reintroduction
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cytosponge-directed Food Reintroduction
Number analyzed (Participants) | 22
score on a scale | 16.5 [9.0 to 28.8]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study for approximately one year on all participants
Arm/Group | Cytosponge-directed Food Reintroduction
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT02599558/Prot_000.pdf